CLINICAL TRIAL: NCT06776055
Title: A Multicenter, Open-label, Long-term Extension Study to Evaluate the Long-term Protective Efficacy and Immunogenic Persistence of the Bivalent Human Papillomavirus Vaccine (Pichia Pastoris) Administered to Healthy Females Aged 18-30 During the 311-HPV-1003 Study
Brief Title: Long-term Follow-up of Bivalent Human Papillomavirus (HPV) Vaccine Study in Women
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai Zerun Biotechnology Co.,Ltd (Industry)
Collaborators: Yuxi Zerun Biotechnology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 311-HPV-1003-EXTEND; 311-HPV-1003-EXTEND (Other: Shanghai Zerun Biotech)
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Cervical Cancer; Vulvar Cancer; Vaginal Cancer; CIN - Cervical Intraepithelial Neoplasia; Human Papillomavirus Infection
Keywords: Bivalent HPV vaccine; Long-term protective efficacy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Uterine Cervical Dysplasia; Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — 1. Cervical Samples:
     Cervical exfoliated cells collected at the 96-month and 120-month visits for ThinPrep Cytologic Testing (TCT) and HPV DNA typing.
  2. Biopsy Samples:
  Tissue samples collected during colposcopy procedures, if biopsy is deemed necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HPV-2 vaccine group: Participants received the bivalent HPV vaccine (0.5 mL in a 3-dose regimen) in the base study (NCT02733068). No study vaccination will be administered in long-term follow-up study .
  Interventions: Biological: HPV-16/18 vaccine
- Placebo group: Participants received the placebo (0.5 mL in a 3-dose regimen) in the base study (NCT02733068). No study vaccination will be administered in long-term follow-up study .
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: HPV-16/18 vaccine — Recombinant human papillomavirus virus-like particle vaccine (Type 16 and 18 L1 Proteins, Yeast)
  Groups: HPV-2 vaccine group
Biological: Placebo — Placebo containing the same formulation as the active vaccine (Type 16 and 18 L1 proteins, Yeast) but without the active substance.
  Groups: Placebo group

SUMMARY:
This extension study aims to evaluate the long-term protection and immune response of the bivalent HPV vaccine in women aged 18-30 who participated in a previous efficacy study (311-HPV-1003). Participants will be monitored over two years, with two visits at 96 and 120 months after their initial vaccination. No additional vaccine doses will be given. Cervical samples will be obtained for ThinPrep Cytologic Testing (TCT) and HPV DNA typing. If applicable, participants meeting referral criteria for colposcopy will undergo the procedure during these visits, and tissue samples will be collected from those requiring a biopsy. Blood samples will be drawn from an immunology subset for antibody testing.The study includes data collection from multiple sites across China to assess the vaccine's long-term efficacy in preventing HPV-related cervical diseases and its durability over time.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to understand and provide informed consent by signing the informed consent form (non-illiterate).
* Have the ability to comply with protocol requirements, such as attending scheduled visits and responding to follow-up phone calls.
* Prior enrollment in the 311-HPV-1003 study, with at least one dose of the study vaccine administered.
* At least one documented gynecological visit between 6 and 48 months during the previous 311-HPV-1003 study.
* Refrain from vaginal intercourse for 48 hours and avoid behaviors such as vaginal douching or using vaginal medications that could interfere with gynecological examinations or sample collection for 72 hours prior to each gynecological visit.

Exclusion Criteria:

* Participants who received another HPV vaccine during the prior 311-HPV-1003 study or between the end of that study and enrollment in this extension study.
* Participants diagnosed with HPV 16- or 18-related CIN2+ by an independent pathology expert panel during the prior 311-HPV-1003 study, or who were definitively diagnosed with HPV 16- or 18-related CIN2+ through external testing after the prior study ended.
* Participants who, at baseline in the 311-HPV-1003 study, tested positive for both HPV 16 and 18 antibodies, or were positive for both HPV 16 and 18 (by Cobas 4800), or whose cytology was not normal or of low-grade changes.
* Participants who are pregnant at the time of gynecological visits or within three months prior to the visit.
* Participants with any other factors deemed unsuitable for participation in the clinical trial, as determined by the investigator.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Participants in this long-term follow-up study were originally enrolled in the 311-HPV-1003 study and are drawn from multiple clinical sites across four provinces in China, including Guangxi, Hebei, Henan, and Shanxi. These participants represent a community-based sample of healthy women who received at least one dose of the Bivalent HPV vaccine or Placebo during the original study.
Sampling Method: Probability Sample
Enrollment: 5372 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Cumulative Protective Efficacy Against HPV-16 and/or HPV-18-Related Cervical Intraepithelial Neoplasia (CIN) Grade 2 or Higher (CIN2+), Adenocarcinoma In Situ (AIS), and Cervical Cancer | Up to 96 months and 120 months after initial vaccination in base study.

SECONDARY OUTCOMES:
Cumulative protective efficacy against cytological HPV-16 and/or HPV-18 infection | Up to 96 months and 120 months after initial vaccination in base study.
Cumulative protective efficacy against HPV-16 and/or HPV-18-related CIN1+ | Up to 96 months and 120 months after initial vaccination in base study.
HPV 16/18 neutralizing antibody GMT and seropositivity rates | At 96 months and 120 months after initial vaccination in base study.

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Lingchuan Center for Disease Control and Prevention, Lingchuan, Guangxi
  - Quanzhou Center for Disease Control and Prevention, Quanzhou, Guangxi
  - Xing'an Center for Disease Control and Prevention, Xing’an, Guangxi
  - Daming Center for Disease Control and Prevention, Daming, Hebei
  - Dingxing Center for Disease Control and Prevention, Dingxing, Hebei
  - Zhengding Center for Disease Control and Prevention, Zhengding, Hebei
  - Puyang Center for Disease Control and Prevention, Puyang, Henan
  - Wenxian Center for Disease Control and Prevention, Wenquan, Henan
  - Xiangfen County People's Hospital, Xincheng, Shanxi